CLINICAL TRIAL: NCT00219635
Title: A Phase 2, Multi-Center, Double-Blind, Placebo-Controlled, Flexible Dose Study To Assess The Efficacy and Safety Of Oral UK-390,957 In Men With Premature Ejaculation
Brief Title: Assessment Of Efficacy and Safety UK-390,957 In Men With Premature Ejaculation
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: A3871029
Record Dates: First submitted 2005-09-09; First posted 2005-09-22 (Estimated); Last update posted 2012-11-07 (Estimated); Status verified 2012-11

CONDITIONS: Ejaculation

INTERVENTIONS:
Drug: UK-390,957

SUMMARY:
Assessment of efficacy and safety UK-390,957

ELIGIBILITY:
Inclusion Criteria:

* Premature ejaculation as defined by DSM-IV

Exclusion Criteria:

* History of erectile dysfunction

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 138
Dates: Start 2005-01; Primary Completion 2005-07 (Actual); Study Completion 2005-07 (Actual)

PRIMARY OUTCOMES:
Assessment of efficacy and safety

SECONDARY OUTCOMES:
Assessment of quality of sexual life

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (22):
- United States (14):
  - Pfizer Investigational Site, Birmingham, Alabama
  - Pfizer Investigational Site, San Bernardino, California
  - Pfizer Investigational Site, Metairie, Louisiana
  - Pfizer Investigational Site, Watertown, Massachusetts
  - Pfizer Investigational Site, Kansas City, Missouri
  - Pfizer Investigational Site, Washington, Missouri
  - Pfizer Investigational Site, New York, New York
  - Pfizer Investigational Site, Williamsville, New York
  - Pfizer Investigational Site, Beachwood, Ohio
  - Pfizer Investigational Site, Portland, Oregon
  - Pfizer Investigational Site, Knoxville, Tennessee
  - Pfizer Investigational Site, Dallas, Texas
  - Pfizer Investigational Site, Houston, Texas
  - Pfizer Investigational Site, Milwaukee, Wisconsin
- Australia (2):
  - Pfizer Investigational Site, St Leonards, New South Wales
  - Pfizer Investigational Site, Malvern, Victoria
- Canada (4):
  - Pfizer Investigational Site, Victoria, British Columbia
  - Pfizer Investigational Site, Barrie, Ontario
  - Pfizer Investigational Site, London, Ontario
  - Pfizer Investigational Site, Toronto, Ontario
- United Kingdom (2):
  - Pfizer Investigational Site, Nr Lichfield, Staffordshire
  - Pfizer Investigational Site, Devon

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A3871029&StudyName=Assessment+Of+Efficacy+and+Safety+UK%2D390%2C957+In+Men+With+Premature+Ejaculation